CLINICAL TRIAL: NCT00230646
Title: Promoting Physical Activity After Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CA101770
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2005-09

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: cancer recovery; physical activity
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Exercise counseling

SUMMARY:
Colorectal cancer is the third most common cancer in the U.S. and if detected early, has a favorable prognosis. Colorectal cancer survivors report increased fatigue, low vigor, impaired physical functioning and disturbances in body esteem. However, the group is relatively understudied and the potential benefits of increased physical activity to their recovery have not been examined. This study focuses on enhancing recovery by offering a home-based physical activity program to patients who have completed treatment for colorectal cancer. This study will test the efficacy of the physical activity intervention using a randomized controlled design among 134 patients who have completed treatment for colorectal cancer in the past 2 years. Outcomes will include physical activity behavior, fitness, vigor, fatigue, physical functioning, and body esteem among participants at baseline, 3 (posttreatment), 6 and 12 months. We will also track intervention costs and conduct exploratory analyses of moderators and mediators of change to help guide the future development of physical activity interventions to enhance recovery from colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer in the U.S. and if detected early, has a favorable prognosis. Colorectal cancer survivors face many physical and psychosocial sequelae including second cancers, adverse effects on major organs, cognitive, and sexual function, problems in work and social roles and reduced quality of life. Following adjuvant treatments (chemotherapy and/or radiation), these individuals may be at increased risk for cardiovascular disease, obesity, osteoporosis and future cancers. There is growing evidence that moderate-intensity physical activity can improve physical functioning, reduce fatigue, enhance vigor and improve body esteem among those treated for breast cancer. Colorectal cancer survivors report increased fatigue, low vigor, impaired physical functioning and disturbances in body esteem. However, the group is relatively understudied and the potential benefits of increased physical activity to their recovery have not been examined. This study focuses on enhancing recovery by offering a home-based physical activity program to patients who have completed treatment for colorectal cancer. The program, based on our prior work among breast cancer survivors, consists of telephone-delivered physical activity counseling over three months. The counseling is based on the Transtheoretical Model, Social Cognitive Theory and elements of Motivational Interviewing. This study will test the efficacy of the physical activity intervention using a randomized controlled design among 134 patients who have completed treatment for colorectal cancer in the past 2 years. Outcomes will include physical activity behavior, fitness, vigor, fatigue, physical functioning, and body esteem among participants at baseline, 3 (posttreatment), 6 and 12 months. We will also track intervention costs and conduct exploratory analyses of moderators and mediators of change to help guide the future development of physical activity interventions to enhance recovery from colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:1) men and women aged >18 years, 2) completed primary and adjuvant treatment for colon or rectal cancer (Stages 1-3). To allow for adequate recovery from treatment, patients whose only treatment is surgery, will be eligible for study participation 12 weeks after surgery and remain eligible for 2 years. Patients who have received chemotherapy or radiation will become eligible 8 weeks after treatment completion, and will remain eligible up to 2 years posttreatment. 3) <2 years since treatment completion, 4) able to read and speak English, 5) provide consent for medical chart review, 6) able to walk unassisted, 7) sedentary which will be defined as: currently not exercising for >30 mins. of moderate-intensity activity on >2 days per week or >20 mins. of vigorous activity one or more days per week over the past 6 months, and 8) have access to a telephone.

-

Exclusion Criteria:Diabetes, hyperlipidemia and uncontrolled hypertension. Patients who have a positive cardiac history (myocardial infarction, angina, peripheral vascular disease, claudication, transient ischemic attacks, claudication, and past history of stroke) will be asked to obtain written permission from their cardiologist prior to study enrollment.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Minutes of moderate-intensity physical activity (PA) at 3 months among 134 sedentary patients who have completed treatment for colorectal cancer (CRC).

SECONDARY OUTCOMES:
Examine the effects of the intervention on survivors' physical functioning, fitness, vigor, fatigue and body esteem at 3 months.
Examine the maintenance of outcomes (minutes of moderate intensity activity, physical functioning, vigor, fatigue and body esteem) at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardine M Pinto, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- Centers for Behavioral and Preventive Medicine, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Kindred MM, Pinto BM, Dunsiger SI. Association of Body Esteem with Fitness and Body Fat Among Colorectal Cancer Survivors: Secondary Analyses from a Randomized Trial. Int J Behav Med. 2019 Dec;26(6):619-628. doi: 10.1007/s12529-019-09819-x. PMID 31650480